CLINICAL TRIAL: NCT01164930
Title: Impact of Acceptance and Commitment Therapy on Salivary Cortisol in Breast Cancer
Brief Title: Impact of Acceptance and Commitment Therapy on Early Stage Breast Cancer
Acronym: ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Jose State University (Other)
Responsible Party: Principal Investigator, Jennifer A. Gregg, PhD, Assistant Professor, San Jose State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5R03CA144751-02 (NIH)
Record Dates: First submitted 2010-07-15; First posted 2010-07-19 (Estimated); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Breast Neoplasms; Survivorship; Stress
MeSH Terms: conditions — Breast Neoplasms | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acceptance and Commitment Therapy group (Experimental): 8-week ACT group
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Wait-list control group (No Intervention): Participants will be offered treatment following wait-list data collection

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — 8-week ACT group
  Arms: Acceptance and Commitment Therapy group

SUMMARY:
The purpose of this randomized controlled trial is to evaluate the effectiveness of an empirically supported psychosocial treatment, Acceptance and Commitment Therapy, in facilitating improved quality of life, benefit-finding, and cortisol rhythm in breast cancer patients in an outpatient clinical oncology setting.

DETAILED DESCRIPTION:
Previous research indicates that breast cancer patients may demonstrate disrupted diurnal cortisol rhythms compared to healthy individuals, and that these disrupted rhythms may be related to recurrence and earlier mortality in some patients. Interestingly, improvements in cortisol regulation in previous intervention studies for cancer patients have not necessarily been related to decreased distress. Rather, improvements in post-traumatic growth, benefit-finding, and meaningfulness have also accounted for improved neuroendocrine and immunological changes.

Traditional breast cancer groups, however, may not adequately address these areas because existing interventions often target the reduction of distress as the primary vehicle to improve psychosocial, quality of life, and biophysical outcomes. Acceptance and Commitment Therapy (ACT) is an empirically-supported, mindfulness-based psychological treatment that has been shown to enhance meaningful behavior change thorough increasing emotional acceptance of difficult psychological experiences such as distress, without the goal of changing or eliminating them.

The current study seeks to determine the preliminary effect of an 8-week ACT group in increasing positive life changes and corresponding increase in salivary cortisol slope in 40 distressed breast cancer patients, who will be randomly assigned to ACT or a wait list control group.

The hypotheses for the present study include:

* Patients receiving ACT will demonstrate improvements in Quality of Life (QoL), Benefit-finding (BF), and health behavior compared to control group participants
* ACT participants will demonstrate improvements in mean cortisol levels and cortisol reactivity compared to control group participants
* These changes will be the result of increased mindful acceptance of cancer-related distress and meaningful behavior changes, rather than a reduction in distress.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of stage I-III breast cancer
* prescreen distress score above defined cutoff
* agreement not to seek other breast cancer support services until study completion

Exclusion Criteria:

* previous cancer
* prior psychiatric treatment for serious mental health disorder (e.g., hospitalization or formal diagnosis of psychosis, major depressive episode, borderline mental retardation, suicidality, or current substance dependence)
* current use of medications known to interfere with cortisol levels (e.g., dexamethasone)
* major concurrent medical disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
salivary cortisol | 3-month follow-up

SECONDARY OUTCOMES:
self-reported distress | 3-month follow-up
self-reported quality of life | 3-month follow-up
self-reported benefit-finding | 3-month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- San Jose State University, San Jose, California, United States